CLINICAL TRIAL: NCT00977912
Title: Prevention of NEC in Preterm Infants With B. Lactis
Brief Title: Necrotizing Enterocolitis (Nec) and B. Lactis in Premature Babies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08.09.INF
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Necrotizing Enterocolitis
Keywords: B. lactis; Preterm; Necrotizing Enterocolitis (NEC)
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Milk" containing B. Lactis (Experimental): "Milk" = Breast-milk from the mother, pasteurized breast-milk from a donor, or preterm formula.
  Interventions: Dietary Supplement: Probiotic supplementation
- "Milk" containing placebo (Placebo Comparator): "Milk" = Breast-milk from the mother, pasteurized breast-milk from a donor, or preterm formula.
  Interventions: Dietary Supplement: Milk containing placebo

INTERVENTIONS:
Dietary Supplement: Probiotic supplementation — one capsule containing probiotics per day added to milk
  Arms: "Milk" containing B. Lactis
Dietary Supplement: Milk containing placebo — one capsule containing placebo per day added to milk
  Arms: "Milk" containing placebo

SUMMARY:
The purpose of the trial is to demonstrate the effect of B. lactis in reducing the incidence of Necrotizing Enterocolitis (NEC) compared to placebo in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 800 - 1500g
* Tolerating enteral feeding within 48 hours
* Having obtained his/her parents or legal representative informed consent

Exclusion Criteria:

* Chromosomal abnormality
* Hydrops featalis
* Congenital malformation of the gastrointestinal tract
* Congenital heart defects or other major congenital abnormalities likely to affect feeding and/or feeding tolerance
* Currently participating in another clinical trial

Ages: 12 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2009-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
NEC onset | 6 weeks

SECONDARY OUTCOMES:
Antibiotic administration and stool microbiology | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Cooper, MD, Principal Investigator — University of Witwatetersrand & Charlotte Maxek Johannestburg Academic Hospital
Locations (3):
- South Africa (3):
  - University of Witwatersrand & Chris Hani Baragwanath Hospital, Bertsham
  - University of Witwatetersrand & Charlotte Maxek Johannestburg Academic Hospital, Johannesburg
  - University of Witwatersrand & Rahima Moosa Mother & Child Hospital, Johannesburg

REFERENCES:
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2023 Jul 26;7(7):CD005496. doi: 10.1002/14651858.CD005496.pub6. PMID 37493095
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2020 Oct 15;10(10):CD005496. doi: 10.1002/14651858.CD005496.pub5. PMID 33058137